CLINICAL TRIAL: NCT04043663
Title: Effects of Virtual Reality on Perioperative Pediatric Anxiety
Acronym: VIRTUALPED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Teresa Franco, Principal investigator, Medical Doctor, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIRTUALPED
Record Dates: First submitted 2019-07-25; First posted 2019-08-02 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Preoperative Anxiety; Maladaptive Postoperative Behavior; Emergence Delirium
Keywords: virtual reality; pediatric surgery
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality program group (Experimental): Virtual reality program based on a virtual reality guided tour registered in the investigator's pediatric OR setting before surgery.
  Interventions: Device: Virtual Reality glasses
- control group (Active Comparator): standard perioperative care without virtual reality program
  Interventions: Procedure: standard perioperative care without virtual reality program

INTERVENTIONS:
Device: Virtual Reality glasses — Children are encouraged to watch the virtual reality program at least 24 hours before surgery.
  Arms: Virtual reality program group
Procedure: standard perioperative care without virtual reality program — standard perioperative care without virtual reality program
  Arms: control group

SUMMARY:
This study evaluates the effect of virtual reality on anxiety levels in a pediatric surgical population. Half of participants will receive standard perioperative treatment, while the other half will receive additionally a virtual reality local program.

DETAILED DESCRIPTION:
It is well known that there is a high incidence of significant anxiety in pediatric population perioperatively, with adverse side effects in terms of emergence delirium and maladaptive postoperative behaviors. Many different strategies have been designed in order to minimize these negative consequences.

Virtual reality is a new and simple technology that can be used at young ages. The aim of this study is to measure anxiety levels at different times in children scheduled for ambulatory surgery compared to patients with standard care without virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* Child between 4 and 12 years old
* Elective ambulatory surgery
* Parents posses a smart phone
* Child and parents understand Spanish or Catalan
* Patient information has been explained
* Informed Consent is signed
* Surgery scheduled in the morning

Exclusion Criteria:

* Child has hearing impairment
* Child has visual impairment
* Child has previous experience of anesthesia
* American Society os Anesthesiologists (ASA) score of III or greater
* Children with history of seizures
* Children under psychiatric treatment

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Perioperative Anxiety level | baseline to 1 day
  In children: measured using the modified Yale Perioperative Anxiety Scale, blinded reported by a trained nurse before the patient is transferred to the operating room. Rage from 23.5 up to 100, deemed high anxiety level if test rated over 30

SECONDARY OUTCOMES:
Salivary Cortisol level | baseline to 1 day
  In children: Saliva sample collection using Salivette system before the patient is transferred to the operating room. Levels over 8nmol/l can be caused by high anxiety level

OTHER OUTCOMES:
Anxiety levels | baseline to 1 day
  In parents: State Anxiety Inventory Scale, self questionnaire made of 20 questions rated from 0 to 3 at the holding area. Range from 1 up to 10

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Franco, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Teresa Franco, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No